CLINICAL TRIAL: NCT03336216
Title: A Phase 2 Study of Cabiralizumab (BMS-986227, FPA008) Administered in Combination With Nivolumab (BMS-936558) With and Without Chemotherapy in Patients With Advanced Pancreatic Cancer
Brief Title: A Study of Cabiralizumab Given With Nivolumab With and Without Chemotherapy in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA025-006
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — cabiralizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; irinotecan sucrosofate; Nivolumab; Fluorouracil; Gemcitabine; Oxaliplatin; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Active Comparator): Investigator choice of chemotherapy:
  Gemcitabine/Nab-Paclitaxel (Abraxane®) or 5-Fluorouracil/Leucovorin/Irinotecan Liposome (ONIVYDE)
  Interventions: Drug: Nab-paclitaxel; Drug: Onivyde; Drug: Fluorouracil; Drug: Gemcitabine; Drug: Leucovorin; Drug: Irinotecan Hydrochloride
- Arm B (Experimental): Cabiralizumab Q2W + Nivolumab Q4W
  Interventions: Biological: Cabiralizumab; Biological: Nivolumab
- Arm C (Experimental): Cabiralizumab Q2W + Nivolumab Q4W and Gemcitabine + Nab-Paclitaxel (Abraxane®) D1, 8 and 15 Q4W
  Interventions: Biological: Cabiralizumab; Drug: Nab-paclitaxel; Biological: Nivolumab; Drug: Gemcitabine
- Arm D (Experimental): Cabiralizumab Q2W + Nivolumab Q4W and Oxaliplatin/5-Flurouracil/Leucovorin (FOLFOX) Q2W
  Interventions: Biological: Cabiralizumab; Biological: Nivolumab; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Biological: Cabiralizumab — specified dose on specified days
  Other Names: BMS-986227, FPA008
  Arms: Arm B; Arm C; Arm D
Drug: Nab-paclitaxel — specified does on specified days
  Other Names: Abraxane
  Arms: Arm A; Arm C
Drug: Onivyde — specified dose on specified days
  Other Names: irinotecan liposome
  Arms: Arm A
Biological: Nivolumab — specified dose on specified days
  Other Names: Opdivo, BMS-936558
  Arms: Arm B; Arm C; Arm D
Drug: Fluorouracil — specified dose on specified days
  Other Names: 5-Fluorouracil
  Arms: Arm A; Arm D
Drug: Gemcitabine — specified dose on specified days
  Arms: Arm A; Arm C
Drug: Oxaliplatin — specified dose on specified day
  Arms: Arm D
Drug: Leucovorin — Specified dose on specified days
  Arms: Arm A; Arm D
Drug: Irinotecan Hydrochloride — Specified dose on specified days
  Arms: Arm A

SUMMARY:
The purpose of this study is to determine whether an investigational immuno-therapy, cabiralizumab in combination with nivolumab, with or without chemotherapy, is effective for the treatment of advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have histological or cytological confirmed diagnosis of locally advanced or metastatic adenocarcinoma of the pancreas, which has progressed on or after one line of chemotherapy
* ECOG Performance status 0-1
* Adequate organ functions
* Measurable disease

Exclusion Criteria:

* Suspected or known CNS metastasis
* Participants with active, known, or suspected autoimmune disease
* Uncontrolled or significant cardiovascular disease
* Prior exposure to selected immune cell-modulating antibody regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (19):
  - Mayo Clinic in Rochester, Minnesota, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Local Institution - 0007, Los Angeles, California
  - University Of Colorado, Aurora, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Local Institution - 0001, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Local Institution - 0010, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Local Institution - 0012, New York, New York
  - Local Institution - 0005, New York, New York
  - Local Institution - 0006, Philadelphia, Pennsylvania
  - Local Institution - 0009, Pittsburgh, Pennsylvania
  - Tennessee Oncology Chattanooga, Nashville, Tennessee
  - Local Institution - 0013, Dallas, Texas
  - Local Institution - 0011, Houston, Texas
  - University Of Washington, Seattle, Washington
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Local Institution - 0037, Kingston, Ontario
  - Local Institution - 0035, Toronto, Ontario
- Local Institution - 0041, Herlev, Denmark
- Germany (4):
  - Local Institution - 0032, Heidelberg
  - Local Institution - 0029, Mannheim
  - Universitaetsklinikum Ulm, Ulm
  - Local Institution - 0030, Würzburg
- Italy (2):
  - Local Institution - 0025, Padua
  - Local Institution - 0026, Roma
- Japan (2):
  - Local Institution - 0023, Kashiwa-shi, Chiba
  - Local Institution - 0022, Chuo-ku, Tokyo
- South Korea (2):
  - Local Institution - 0018, Seoul
  - Local Institution - 0017, Seoul
- Spain (3):
  - Local Institution - 0021, Barcelona
  - Local Institution - 0019, Madrid
  - Local Institution - 0020, Madrid
- Switzerland (2):
  - Local Institution - 0033, Chur
  - Local Institution - 0034, Lausanne
- Taiwan (2):
  - Local Institution - 0024, Taipei
  - Local Institution - 0031, Taipei
- Local Institution - 0016, Glasgow, Lanarkshire, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Investigator Choice: Participants receive Investigator choice of chemotherapy:
  * gemcitabine + nab-paclitaxel
  * 5-Fluorouracil/Leucovorin/Irinotecan Liposome
- Arm B: Cabiralizumab + Nivolumab: Participants receive Cabiralizumab 4MG/KG Q2W + Nivolumab 480 MG Q4W.
- Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy: Participants receive Cabiralizumab 4MG/KG Q2W + Nivolumab 480 MG Q4W and Gemcitabine + Nab-paclitaxel D1, 8, and 15 Q4W.
- Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy: Participants receive Cabiralizumab 4MG/KG Q2W + Nivolumab 480 MG Q4W and Oxaliplatin/5-Fluorouracil/Leucovorin Q2W.
Period: Randomization
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Started | 54 | 54 | 54 | 43
Completed | 40 | 49 | 48 | 42
Not Completed | 14 | 5 | 6 | 1
Not completed — Not reported | 2 | 0 | 1 | 0
Not completed — Other reasons | 1 | 1 | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 2 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Participant withdrew consent | 9 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Period: Treatment
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Started | 40 | 49 | 48 | 42
Completed | 0 | 1 | 0 | 1
Not Completed | 40 | 48 | 48 | 41
Not completed — Adverse Event | 2 | 3 | 4 | 4
Not completed — Participant request to discontinue treatment | 2 | 1 | 2 | 2
Not completed — Participant withdrew consent | 7 | 2 | 3 | 2
Not completed — Death | 2 | 3 | 3 | 4
Not completed — Participant no longer meets study criteria | 0 | 1 | 0 | 0
Not completed — Other reasons | 2 | 0 | 0 | 3
Not completed — Disease progression | 23 | 34 | 33 | 26
Not completed — Study drug toxicity | 0 | 3 | 2 | 0
Not completed — Adverse Event unrelated to study drug | 1 | 1 | 1 | 0
Not completed — Disease Recurrence | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy | Total
Number analyzed (Participants) | 54 | 54 | 54 | 43 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (8.6) | 64.2 (9.1) | 59.1 (9.7) | 64.2 (9.6) | 62.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 26 | 26 | 106
  Male | 28 | 26 | 28 | 17 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 1 | 0 | 6
  Not Hispanic or Latino | 46 | 48 | 45 | 41 | 180
  Unknown or Not Reported | 3 | 6 | 8 | 2 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 8 | 8 | 12 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 1 | 3 | 12
  White | 40 | 43 | 45 | 27 | 155
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by BICR
Description: PFS for a participant is defined as the time from randomization date to the date of first objectively documented disease progression by blinded independent central review (BICR) per response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Based on Kaplan-Meier Estimates.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization date to the date of first objectively documented disease progression or death (up to approximately 65 months)
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Months | 3.52 [2.53 to 4.21] | 1.92 [1.77 to 2.14] | 3.68 [1.94 to 4.83] | 3.22 [2.04 to 3.94]
Statistical Analysis 1: Comparison: Arm A: Investigator Choice vs Arm B: Cabiralizumab + Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.47, 60% CI 2-sided [1.19 to 1.82]
Statistical Analysis 2: Comparison: Arm A: Investigator Choice vs Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.00, 60% CI 2-sided [0.77 to 1.30]
Statistical Analysis 3: Comparison: Arm A: Investigator Choice vs Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.78, 60% CI 2-sided [0.60 to 1.03]

2. Secondary Outcome: Progression Free Survival (PFS) by Investigator
Description: PFS for a participant is defined as the time from randomization date to the date of first objectively documented disease progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Based on Kaplan-Meier Estimates.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Months | 3.38 [1.97 to 3.98] | 1.81 [1.74 to 1.97] | 3.68 [2.00 to 4.17] | 2.92 [1.81 to 3.94]
Statistical Analysis 1: Comparison: Arm A: Investigator Choice vs Arm B: Cabiralizumab + Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.64, 60% CI 2-sided [1.33 to 2.02]
Statistical Analysis 2: Comparison: Arm A: Investigator Choice vs Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 1.13, 60% CI [0.87 to 1.46]
Statistical Analysis 3: Comparison: Arm A: Investigator Choice vs Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.72, 60% CI [0.55 to 0.94]

3. Secondary Outcome: Progression Free Survival Rate (PFSR) by BICR
Description: Progression Free Survival Rates at 6, 9, and 12 months is defined as the percentage of participants who achieve PFS at 6, 9, and 12 months. PFS for a participant is defined as the time from randomization date to the date of first objectively documented disease progression by blinded independent central review (BICR) per response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Based on Kaplan-Meier Estimates.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: At 6, 9, and 12 months
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Percentage of participants
  6-MONTH | 15.5 [4.8 to 31.8] | 13.1 [5.3 to 24.4] | 21.7 [10.5 to 35.4] | 17.7 [7.8 to 30.8]
  9-MONTH | 5.2 [0.4 to 20.3] | 6.5 [1.7 to 16.1] | 9.5 [2.6 to 21.8] | 10.1 [3.2 to 21.7]
  12-MONTH | NA [NA to NA] — Insufficient number of participants with events | 2.2 [0.2 to 10.0] | 3.2 [0.3 to 13.6] | 5.1 [0.9 to 15.0]

4. Secondary Outcome: Progression Free Survival Rate (PFSR) by Investigator
Description: Progression Free Survival Rates at 6, 9, and 12 months is defined as the percentage of participants who achieve PFS at 6, 9, and 12 months. PFS for a participant is defined as the time from randomization date to the date of first objectively documented disease progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Based on Kaplan-Meier Estimates.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: At 6, 9, and 12 months
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Percentage of participants
  6-MONTH | 14.9 [4.9 to 30.0] | 16.3 [7.6 to 27.9] | 17.6 [8.2 to 29.8] | 14.7 [6.0 to 27.1]
  9-MONTH | 11.2 [3.0 to 25.6] | 8.2 [2.6 to 17.9] | 5.0 [0.9 to 14.7] | 7.3 [1.9 to 17.9]
  12-MONTH | 3.7 [0.3 to 15.9] | NA [NA to NA] — Insufficient number of participants with events | 2.5 [0.2 to 11.2] | 4.9 [0.9 to 14.5]

5. Secondary Outcome: Objective Response Rate (ORR) by BICR
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is either CR or PR by blinded independent central review (BICR) per response evaluation criteria in solid tumors (RECIST) v1.1 based on Clopper-Pearson method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization to the date of objectively documented progression per RECIST v1.1 or the date of subsequent anti-cancer therapy, whichever occurs first (up to approximately 65 months)
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Percentage of participants | 2.5 [0.1 to 13.2] | 4.1 [0.5 to 14.0] | 12.5 [4.7 to 25.2] | 9.5 [2.7 to 22.6]
Statistical Analysis 1: Comparison: Arm A: Investigator Choice vs Arm B: Cabiralizumab + Nivolumab; Test type: Superiority; p = 0.6537, Cochran-Mantel-Haenszel — Stratified CMH test stratified by ECOG and prior chemotherapy; Strata adjusted difference = 1.8, 95% CI [-5.5 to 9.0] — Based on Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 2: Comparison: Arm A: Investigator Choice vs Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy; Test type: Superiority; p = 0.0951, Cochran-Mantel-Haenszel — Stratified CMH test stratified by ECOG and prior chemotherapy; Strata adjusted difference = 12.5, 95% CI [3.1 to 21.9] — Based on Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 3: Comparison: Arm A: Investigator Choice vs Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy; Test type: Superiority; p = 0.5171, Cochran-Mantel-Haenszel — Stratified CMH test stratified by ECOG and prior chemotherapy; Strata adjusted difference = 5.0, 95% CI [-8.0 to 18.1] — Based on Cochran-Mantel-Haenszel (CMH) method of weighting

6. Secondary Outcome: Objective Response Rate (ORR) by Investigator
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is either CR or PR per response evaluation criteria in solid tumors (RECIST) v1.1 based on Clopper-Pearson method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 5
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Percentage of participants | 5.0 [0.6 to 16.9] | 4.1 [0.5 to 14.0] | 6.3 [1.3 to 17.2] | 4.8 [0.6 to 16.2]
Statistical Analysis 1: Comparison: Arm A: Investigator Choice vs Arm B: Cabiralizumab + Nivolumab; Test type: Superiority; p = 0.8505, Cochran-Mantel-Haenszel — Stratified CMH test stratified by ECOG and prior chemotherapy; Strata adjusted difference = -0.8, 95% CI 2-sided [-9.4 to 7.7] — Based on Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 2: Comparison: Arm A: Investigator Choice vs Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy; Test type: Superiority; p = 0.8144, Cochran-Mantel-Haenszel — Stratified CMH test stratified by ECOG and prior chemotherapy; Strata adjusted difference = 1.5, 95% CI 2-sided [-9.9 to 12.8] — Based on Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 3: Comparison: Arm A: Investigator Choice vs Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy; Test type: Superiority; p = 0.9087, Cochran-Mantel-Haenszel — Stratified CMH test stratified by ECOG and prior chemotherapy; Strata adjusted difference = 0.7, 95% CI 2-sided [-10.7 to 12.1] — Based on Cochran-Mantel-Haenszel (CMH) method of weighting

7. Secondary Outcome: Duration of Response (DOR) by BICR
Description: DOR for a participant with a best overall response (BOR) of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression by blinded independent central review (BICR) per response evaluation criteria in solid tumors (RECIST) v1.1 or death, whichever occurs first. Median computed using Kaplan-Meier method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization the date of the first objectively documented tumor progression or death, whichever occurs first (up to approximately 65 months)
Population: All Confirmed Responders: All efficacy evaluable participants (randomized population with at least one dose of study drug) with CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 1 | 2 | 6 | 4
Months | NA [NA to NA] — Insufficient number of participants with events. | 4.2 [3.9 to NA] — Insufficient number of participants with events. | 4.6 [3.0 to NA] — Insufficient number of participants with events. | NA [5.6 to NA] — Insufficient number of participants with events.

8. Secondary Outcome: Duration of Response (DOR) by Investigator
Description: DOR for a participant with a best overall response (BOR) of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death, whichever occurs first. Median computed using Kaplan-Meier method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 2 | 2 | 3 | 2
Months | 10.2 [2.7 to NA] — Insufficient number of participants with events. | 7.3 [4.5 to NA] — Insufficient number of participants with events. | NA [3.7 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death due to any cause. Based on Kaplan-Meier Estimates.
Time Frame: From randomization to the date of death to any cause (up to approximately 65 months)
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Months | 6.28 [4.53 to 8.11] | 4.44 [3.19 to 7.26] | 6.72 [4.96 to 8.54] | 5.68 [4.57 to 7.33]
Statistical Analysis 1: Comparison: Arm A: Investigator Choice vs Arm B: Cabiralizumab + Nivolumab; Test type: Superiority; Cox Proportional Hazard = 1.22, 95% CI 2-sided [0.76 to 1.96] — Stratified Cox proportional hazard model by ECOG and type of prior chemotherapy
Statistical Analysis 2: Comparison: Arm A: Investigator Choice vs Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy; Test type: Superiority; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.59 to 1.86] — Stratified Cox proportional hazard model by ECOG and type of prior chemotherapy
Statistical Analysis 3: Comparison: Arm A: Investigator Choice vs Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy; Test type: Superiority; Cox Proportional Hazard = 0.81, 95% CI 2-sided [0.45 to 1.46] — Stratified Cox proportional hazard model by ECOG and type of prior chemotherapy

10. Secondary Outcome: Overall Survival Rates (OSR)
Description: Overall survival at 6 months, 1 year, and 2 years is defined as the percentage of participants who are alive at 6 months, 1 year, and 2 years. Based on Kaplan-Meier Estimates.
Time Frame: At 6 months, 1 year, and 2 years
Population: All Efficacy Participants: Randomized population with at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Percentage of participants
  6-MONTH | 55.8 [38.8 to 69.8] | 40.1 [26.1 to 53.8] | 54.2 [39.2 to 67.0] | 44.8 [29.4 to 59.0]
  12-MONTH | 14.7 [5.4 to 28.3] | 20.1 [10.0 to 32.7] | 20.6 [10.6 to 33.0] | 17.4 [7.7 to 30.4]
  24-MONTH | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

11. Secondary Outcome: The Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 51 months)
Population: All treated participants: All participants who take at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Participants | 40 | 49 | 48 | 42

12. Secondary Outcome: The Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 51 months)
Population: All treated participants: All participants who take at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Participants | 23 | 41 | 39 | 33

13. Secondary Outcome: The Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 11
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 51 months)
Population: All treated participants: All participants who take at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Participants | 6 | 11 | 11 | 8

14. Secondary Outcome: The Number of Participants Who Died
Description: The number of participants that died during the study.
Time Frame: From first dose to 150 days after last dose of study therapy (up to approximately 53 months)
Population: All treated participants: All participants who take at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 40 | 49 | 48 | 42
Participants | 25 | 33 | 30 | 28

15. Secondary Outcome: The Number of Participants Who Experienced Abnormal Hepatic Tests
Description: The number of treated participants who experienced a laboratory abnormality of the liver during the course of the study.
  Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Upper Limit of Normal (ULN)
Time Frame: From first dose and 100 days after last dose of study therapy (up to approximately 51 months)
Population: All treated participants with at least one on-treatment hepatic measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 38 | 45 | 45 | 41
Participants
  ALT or AST > 3xULN | 2 | 21 | 37 | 34
  ALT or AST > 5xULN | 0 | 10 | 19 | 18
  ALT or AST > 10xULN | 0 | 2 | 6 | 2
  ALT or AST > 12xULN | 0 | 2 | 4 | 2
  ALT or AST > 20xULN | 0 | 1 | 1 | 1
  TOTAL BILIRUBIN > 2xULN | 3 | 3 | 2 | 5
  ALP > 1.5xULN | 27 | 31 | 35 | 30
  ALT/AST > 3xULN; TOTAL BILIRUBIN > 2xULN and ALP <=2ULN IN 3 DAYS | 0 | 1 | 1 | 1

16. Secondary Outcome: The Number of Participants With On-Treatment Laboratory Abnormalities in Specific Thyroid Tests
Description: The number of treated participants who experienced a laboratory abnormality of the thyroid during the course of the study.
  Free T3 (FT3) Free T4 (FT4) Lower Limit of Normal (LLN) Upper Limit of Normal (ULN)
Time Frame: From first dose and 100 days after last dose of study therapy (up to approximately 51 months)
Population: All treated participants with at least one on-treatment thyroid stimulating hormone (TSH) measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Investigator Choice | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
Number analyzed (Participants) | 11 | 23 | 25 | 20
Participants
  TSH > ULN | 3 | 4 | 10 | 6
  TSH > ULN WITH TSH <= ULN AT BASELINE | 0 | 2 | 4 | 2
  TSH > ULN WITH AT LEAST ONE T3/T4 TEST VALUE < LLN | 0 | 1 | 1 | 0
  TSH > ULN WITH ALL T3/T4 TEST VALUES >= LLN | 0 | 0 | 0 | 0
  TSH > ULN WITH T3/T4 TEST MISSING | 0 | 1 | 0 | 0
  TSH < LLN | 0 | 0 | 1 | 1
  TSH < LLN WITH TSH >= LLN AT BASELINE | 0 | 0 | 0 | 1
  TSH < LLN WITH AT LEAST ONE T3/T4 TEST VALUE > ULN | 0 | 0 | 0 | 0
  TSH < LLN WITH ALL OTHER T3/T4 TEST VALUES <= ULN | 0 | 0 | 0 | 0
  TSH < LLN WITH T3/T4 TEST MISSING | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from a participants first dose to their study completion (up to approximately 65 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 51 months)
Description: The number at Risk for All-Cause Mortality represents all randomized participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Arm A1: Investigator Choice - Gem/Nab-Based Chemotherapy: Participants receive Investigator choice of chemotherapy:
  - gemcitabine + nab-paclitaxel
- Arm A2: Investigator Choice - 5 FU-Based Chemotherapy: Participants receive Investigator choice of chemotherapy:
  - 5-Fluorouracil/Leucovorin/Irinotecan Liposome
Arm/Group | Arm A1: Investigator Choice - Gem/Nab-Based Chemotherapy | Arm A2: Investigator Choice - 5 FU-Based Chemotherapy | Arm B: Cabiralizumab + Nivolumab | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy
All-Cause Mortality (participants affected / at risk) | 19/26 | 17/28 | 49/54 | 49/54 | 40/43
Serious Adverse Events (participants affected / at risk) | 11/21 | 12/19 | 41/49 | 39/48 | 33/42
Other Adverse Events (participants affected / at risk) | 19/21 | 17/19 | 46/49 | 47/48 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Investigator Choice - Gem/Nab-Based Chemotherapy (N=21) | Arm A2: Investigator Choice - 5 FU-Based Chemotherapy (N=19) | Arm B: Cabiralizumab + Nivolumab (N=49) | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy (N=48) | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 3 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 3 | 5
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 1 | 2 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 3 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 3 | 4 | 6
Septic shock (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood electrolytes abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 1 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 6 | 22 | 19 | 15
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 4 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Investigator Choice - Gem/Nab-Based Chemotherapy (N=21) | Arm A2: Investigator Choice - 5 FU-Based Chemotherapy (N=19) | Arm B: Cabiralizumab + Nivolumab (N=49) | Arm C: Cabiralizumab + Nivolumab + Gemcitabine-Based Chemotherapy (N=48) | Arm D: Cabiralizumab + Nivolumab + 5-FU-Based Chemotherapy (N=42)
Anaemia (Blood and lymphatic system disorders) | 9 | 5 | 13 | 34 | 17
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 13 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 19 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 3 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 2 | 5 | 1
Halo vision (Eye disorders) | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 13 | 21 | 16
Vision blurred (Eye disorders) | 0 | 0 | 1 | 4 | 3
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 4 | 15 | 7 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 6
Ascites (Gastrointestinal disorders) | 0 | 0 | 4 | 4 | 1
Constipation (Gastrointestinal disorders) | 7 | 8 | 13 | 13 | 12
Defaecation urgency (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 11 | 16 | 24
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 5 | 4 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 6 | 2 | 3
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4 | 3 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 2
Lip dry (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 9 | 19 | 16 | 23
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 2 | 4 | 7 | 13
Vomiting (Gastrointestinal disorders) | 9 | 7 | 11 | 15 | 13
Asthenia (General disorders) | 3 | 1 | 3 | 5 | 5
Catheter site phlebitis (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 5 | 2 | 2 | 8 | 6
Face oedema (General disorders) | 0 | 0 | 3 | 5 | 13
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 10 | 10 | 25 | 29 | 23
Generalised oedema (General disorders) | 0 | 0 | 0 | 5 | 3
Influenza like illness (General disorders) | 1 | 0 | 1 | 5 | 1
Mucosal inflammation (General disorders) | 2 | 2 | 0 | 7 | 7
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 0 | 4 | 15 | 6
Pain (General disorders) | 3 | 0 | 4 | 2 | 1
Peripheral swelling (General disorders) | 2 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 6 | 3 | 12 | 18 | 15
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0 | 3
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 2 | 4 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 5 | 3 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 5 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 9 | 18 | 16
Amylase increased (Investigations) | 0 | 0 | 0 | 4 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 14 | 27 | 24
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 9 | 14 | 10
Blood bilirubin increased (Investigations) | 0 | 0 | 5 | 3 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 15 | 18 | 23
Blood creatinine increased (Investigations) | 1 | 0 | 4 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 7 | 8 | 10
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 1 | 3 | 4 | 6 | 7
Neutrophil count decreased (Investigations) | 7 | 4 | 1 | 6 | 9
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 7 | 3 | 1 | 18 | 8
Weight decreased (Investigations) | 3 | 2 | 5 | 7 | 4
White blood cell count decreased (Investigations) | 4 | 3 | 2 | 11 | 6
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 6 | 11 | 17 | 23
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 9 | 4 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 7 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 7 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 6 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8 | 8 | 9 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 7 | 3 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 5 | 9 | 11
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 9 | 5 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 5 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 5 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 3 | 6 | 7
Dysgeusia (Nervous system disorders) | 1 | 2 | 4 | 4 | 8
Headache (Nervous system disorders) | 1 | 3 | 6 | 5 | 4
Neuropathy peripheral (Nervous system disorders) | 6 | 1 | 0 | 13 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 6 | 9
Polyneuropathy (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 2 | 2
Depression (Psychiatric disorders) | 0 | 0 | 3 | 6 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 7 | 3 | 6
Somnambulism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 4 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 4 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 9 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 5 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 2 | 5 | 13 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 8 | 12 | 6
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 11 | 14 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 7 | 11 | 5
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 2 | 2
Hot flush (Vascular disorders) | 0 | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 8 | 8 | 6
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03336216/Prot_SAP_000.pdf